CLINICAL TRIAL: NCT04478253
Title: Effect of the Use of HYPNO VR on Pain Experienced During Chest Drain Insertion in Resuscitation Vigilant Patients.
Brief Title: Virtual Reality Hypnosis for Thoracic Drain Insertion
Acronym: VeRHiTY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-A02677-50
Record Dates: First submitted 2020-07-02; First posted 2020-07-20 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Pneumopathy
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: Randomized prospective monocentric open-label study on two parallel groups based on the use or non-use of a virtual reality device coupled with hypnosis software (HYPNO-VR) during the insertion of a chest tube.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HypnoVR (Experimental): Insertion of the drain according to the usual management protocol supplemented by the use of a hypnosis software application (HYPNO-VR).
  Interventions: Device: HypnoVR
- Usual care (No Intervention): Insertion of the drain according to the usual management protocol

INTERVENTIONS:
Device: HypnoVR — Insertion of the drain according to the usual management protocol supplemented by the use of a hypnosis software application (HYPNO-VR).
  Arms: HypnoVR

SUMMARY:
The main objective of this study is to evaluate, in vigilant resuscitation patients, the effect of the use of HYPNO VR on the pain felt during the insertion of a thoracic drain.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, monocentric, prospective study of two parallel groups of patients in whom a chest tube is to be inserted:

* Group 1: Insertion of the drain according to the usual management protocol.
* Group 2: Insertion of the drain according to the usual management protocol supplemented by the use of a hypnosis software application (HYPNO-VR).

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older, having read and signed the consent form for participation in the study
* Patient admitted to intensive care whose state of health requires the insertion of a thoracic drain according to the doctor in charge of the patient.

Exclusion Criteria:

* Patient under legal protection, guardianship or trusteeship
* Pregnant or breastfeeding patient
* Patient not affiliated to the French social security system
* Hearing or visual disturbances contraindicating the use of virtual reality headphones
* Inability to provide the subject with informed information and/or written informed consent: dementia, psychosis, consciousness disorders, non-French speaking patient
* Unbalanced epilepsy
* Contraindication to local anaesthesia, one of the analgesics or sleeping pills used in the protocol
* Need for drainage in a life-threatening emergency (respiratory distress or compressive pleural effusion)
* Concurrent participation in other research or during a period of exclusion from previous research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Pain intensity progression | 24 hours
  The intensity of pain associated with chest drain insertion (difference between pain felt at the time of insertion and basal pain prior to the procedure) is the primary endpoint. This will be measured on a simple numerical scale Graduated from 0 (no pain) to 10 (worst pain imaginable). Basal pain will be assessed 15 min before drainage, then immediately after insertion and after 4h, 8h, 12h, 16h, 20h and 24h.

SECONDARY OUTCOMES:
Evolution of pain measured on a simple numerical scale over 24 hours | 24 hours
  Evolution of pain over 24 hours measured on a simple numerical scale Graduated from 0 (no pain) to 10 (worst pain imaginable). Basal pain will be assessed 15 min before drainage, then immediately after insertion and after 4h, 8h, 12h, 16h, 20h and 24h.
Pain distress measured on a simple numerical scale during the procedure and evolution from basal state | 24 hours
  Pain distress during the procedure and evolution from basal state. The patient will rate how much pain during the procedure was distressing or annoying on a simple numerical scale ranging from 0 (not at all) to 10 (very annoying or upsetting). It will be evaluated in the basal state 15 min before drainage, then immediately after insertion and after 24 hours.
Anxiety level measured on a simple numerical scale and the State-trait Anxiety Inventory scale (STAI-Y scale) during the procedure and evolution from basal status | 24 hours
  Anxiety level measured on a simple numerical scale graduated from 0 (no anxiety) to 10 (worst imaginable anxiety) and the State-trait Anxiety Inventory scale (STAI-Y scale) during the procedure and evolution from basal status. The simple numerical scale graded from 0 (no anxiety) to 10 (worst imaginable anxiety) will be evaluated in the basal state 15 min before drainage, then immediately after insertion and after 4h, 8h, 12h, 16h, 20h and 24h. The STAI-Y scale has 20 items evaluated from 1 to 4 according to its intensity (1= NO, 2 = rather NO, 3 = rather YES, 4 = YES) will be evaluated in the basal state 15 min before drainage then immediately after insertion and after 24 hours.
Evaluation of sleep quality simple numerical scale graduated from 0 (very bad) to 10 (very good) on the first night after insertion of the drain and evolution compared to usual sleep quality. | 24 hours
  Evaluation of sleep quality measured on a simple numerical scale graduated from 0 (very bad) to 10 (very good) on the first night after insertion of the drain and evolution compared to usual sleep quality.
Drug consumption during the 24 hours following the insertion of the drain: analgesics (paracetamol, Tramadol, Nefopam, Morphine), Bromazepam and Zopiclone. | 24 hours
  Drug consumption during the 24 hours following the insertion of the drain: analgesics (paracetamol, Tramadol, Nefopam, Morphine), Bromazepam and Zopiclone.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud GALBOIS, MD, Principal Investigator — Hôpital Privé Claude Galien
Locations (1):
- Hôpital Privé Claude Galien, Quincy-sous-Sénart, France